CLINICAL TRIAL: NCT00564031
Title: Hormonal Replacement Therapy and Small Artery Function
Acronym: HRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 166/99; 166/99
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Menopause
Keywords: hormone replacement therapy; endothelial function;
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: Femanest
- 3 (Experimental)
  Interventions: Drug: gestapuran
- 4 (Experimental)
  Interventions: Drug: Femanest plus Gestapuran

INTERVENTIONS:
Drug: Femanest — 2mg/day
  Arms: 2
Drug: gestapuran — 5mg/day
  Arms: 3
Drug: placebo — daily
  Arms: 1
Drug: Femanest plus Gestapuran — combined daily
  Arms: 4

SUMMARY:
Endothelial dysfunction in resistance arteries in women after the menopause is important for the development of high blood pressure and cardiovascular disease

DETAILED DESCRIPTION:
We aim to study the effects of different hormone replacement therapies (HRT) on the function and morphology of resistance arteries, and to look for their mechanistic basis. We expect that HRT with estrogens or in combination with MPA may benefit the function of resistance arteries and may preserve the morphological integrity of endothelial cells by regulatory actions on the cytoskeleton.

ELIGIBILITY:
Inclusion Criteria:

* All women had been amenorrheic for at least 1.5 year.
* Menopausal status was confirmed by a serum concentration of follicular- stimulating hormone (FSH > 34 IU/ml) and estradiol (E2 <50 pmol/l).

Exclusion Criteria:

* Cigarette smokers and women with:

  * Hypertension
  * Diabetes mellitus
  * Clinical manifestations of arteriosclerosis (coronary heart disease, peripheral artery disease, or cerebrovascular disease)
  * Venous thromboembolic disease
  * Liver disorders
  * Unexplained vaginal bleeding; and
  * Personal or family history of breast cancer were excluded.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2003-01; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
endothelium-dependent dilatation | 3 month

SECONDARY OUTCOMES:
pressure-induced tone and vascular morphology | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Kublickiene, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University hospital-huddinge, Stockholm, Sweden